CLINICAL TRIAL: NCT03366051
Title: Sentinel Node Mapping Versus Sentinel Node Mapping With Systematic Lymphadenectomy in High Risk Endometrial Cancer: a Open Label, Non-inferiority, Randomized Trial.
Brief Title: Sentinel Node Mapping in High Risk Endometrial Cancer
Acronym: ALICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Glauco Baiocchi Neto, Director, Department of Gynecologic Oncology, AC Camargo Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.392.088
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Cancer; Lymph Node Metastases
Keywords: Endometrial Cancer; Sentinel Lymph Node; Lymphadenectomy
MeSH Terms: conditions — Endometrial Neoplasms; Lymphatic Metastasis | interventions — Lymph Node Excision

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Non-Inferiority Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sentinel Node Mapping plus Lymphadenectomy (Active Comparator): Patients with high risk endometrial cancer will undergo Sentinel Node Mapping followed by Systematic Pelvic and Para-Aortic Lymphadenectomy
  Interventions: Procedure: Sentinel Node Mapping; Procedure: Lymphadenectomy
- Sentinel Node Mapping (Experimental): Patients with high risk endometrial cancer will undergo Sentinel Node Mapping per NCCN algorithm
  Interventions: Procedure: Sentinel Node Mapping

INTERVENTIONS:
Procedure: Sentinel Node Mapping — At least one sentinel node should be retrieved in both hemipelvis. If no sentinel node is found in one hemipelvis, a side specific lymphadenectomy will be performed.
Procedure: Lymphadenectomy — Systematic Pelvic and Para-Aortic Lymphadenectomy
  Arms: Sentinel Node Mapping plus Lymphadenectomy

SUMMARY:
This study will evaluate the role of systematic lymphadenectomy after sentinel node (SLN) mapping in high risk endometrial cancer (high grade histologies or deep myometrial invasion). The participants will be randomized in a non-inferiority controlled trial in 2 groups: SLN mapping or SLN mapping followed by systematic lymphadenectomy.

DETAILED DESCRIPTION:
Although most patients with endometrial cancer present with early-stage disease, the standard treatment still includes systematic lymph node dissection for staging. Recently, SLN mapping has emerged as an acceptable surgical strategy when deciding between complete lymphadenectomy and no node dissection. This approach can help avoid the morbidity that is associated with a complete lymphadenectomy, such as neurovascular injury, lymphocyst formation, and lymphedema. A recent meta-analysis that included 55 studies and 4915 patients reported an overall SLN detection rate of 81% versus 50% for bilateral SLNs. Moreover, the use of indocyanine green increased the bilateral SLN detection rate compared with blue dye (74.6% vs. 50.5%). Yet, the studies noted an overall sensitivity of 96% and false negative rates of less than 5% when analyzed per hemipelvis. Since 2014, the National Comprehensive Cancer Network (NCCN) guidelines have recommended SLN mapping as an alternative option for node staging in endometrial cancer. However, most studies on SLN mapping have included patients who are at low risk for lymph node involvement and thus might underestimate the false negative rate. Recently, Soliman et al. reported a series of only high-grade and deep invasive endometrial cancers for which patients underwent SLN mapping, followed by pelvic and para-aortic lymph node dissection. An 89% detection rate was reported, suggesting that SLN mapping accurately identifies node metastases, with an negative predictive value (NPV) of 98% and an false negative predictive value (FNPV) of 2% when analyzed by hemipelvises. Positive nodes were found in 22.8% of patients (43% of isolated tumor cells and micrometastases), and in 40% of cases, the SLN was the only positive node. Data from the investigators corroborate these findings-26.7% of high-risk cases had positive nodes (50% of isolated tumor cells and micrometastases), and when analyzed by hemipelvis, the NPV was 97.9% and the FNPV was 2.1%. In 14 (70%) patients, the SLN was the only positive node. Moreover, there are few publications that have compared the results of the addition of SLN mapping to lymphadenectomy alone. Raimond et al. compared 156 patients that had SLN mapping with 95 who had pelvic node dissection. In their study, SLN mapping and imuno-histochemistry (IHC) were performed in low- and intermediate-risk patients, and the former detected metastatic node 3 times more often than complete pelvic lymphadenectomy alone (16.2% vs. 5.1%, p=0.03). They had no false negatives, and the IHC findings modified the adjuvant therapy in half of all cases. Holloway et al. compared a series of 661 patients who had undergone pelvic and para-aortic lymphadenectomy with 119 who were subjected to SLN mapping plus node dissection, including 68 high-intermediate- and high-risk patients in the SLN mapping group (GOG99 stratification). Despite the similarity in demographics and pathological risk factors, the SLN group had more LN metastases that were detected (30.3% vs. 16.3%; p<0.001) and received more adjuvant therapy (28.6% vs. 16.3%; p=0.003). The SLN was the only positive node in 18 (50%) of mapped cases, and the false negative rate was 2.8%.The investigators recently published a series on high risk endometrial cancer and also recorded a higher pelvic node metastasis rate for the SLN mapping group (26.7% vs. 14.3%, p=0.02) but no significant difference in para-aortic node metastases (13.5% vs. 5.6%, p=0.12). Notably, if considered only patients in whom SLNs were mapped, 31.3% had pelvic positive nodes. Despite the differences in uterine risk factors between groups, 10.6% (8/75) of patients in the SLN group had node metastasis that was diagnosed only after IHC. Excluding these patients, the SLN group would have had a node positivity rate of 17.3%, similar to the N-SLN group (17.4%), reinforcing the impact of IHC in the detection of node metastases. Moreover, the SLN group received more adjuvant chemotherapy (33.5% vs. 48%). The overall detection rate for SLNs was 85.3%, and bilateral SLNs were observed in 60%. The investigators noted an overall sensitivity of 90%, a negative predictive value of 95.7%, and a false negative predictive value of 4.3%. Recently, Touhami et al. showed that the risk of non-SLN metastasis is 61% when the SLN metastasis size is ≥2mm, and 5% for SLN metastasis of <2mm. However, one of the remaining uncertainties is the role of systematic lymphadenectomy after a positive SLN. In other words, is there any benefit in favor of systematic lymphadenectomy in a patient that already undergo adjuvant chemotherapy? The investigators hypothesized that there is no disease free survival benefit in adding systematic lymphadenectomy to only sentinel node mapping and proposed a prospective randomized controlled non-inferiority trial comparing SLN mapping to SLN mapping with systematic lymphadenectomy in high risk endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* High grade histologies (endometrioid grade 3, serous, clear cell and carcinosarcoma)
* Endometrioid grades 1 or 2 with myometrial invasion of ≥50%
* Endometrioid grades 1 or 2 with cervical invasion
* Clinically suitable to receive systematic lymphadenectomy
* Consent statement

Exclusion Criteria:

* Previous hysterectomy in other institution
* Presence of extra-uterine disease (peritoneal, visceral or suspicious lymph node metastasis)
* Previous pelvic node dissection

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 3 years
  Recurrence Free Survival

SECONDARY OUTCOMES:
Survival | 5 years
  Overall Survival
Early morbidity | <30 days after surgery
  Surgical and clinical morbidity
Late morbidity | >30 days after surgery
  Surgical and clinical morbidity
Lymphedema | Evaluation before surgery and after 6 and 12 months of follow-up
  Presence and lymphedema graduation
Quality of Life Questionary (QLQ) | Evaluation before surgery and after 1 and 6 months of follow-up
  EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Glauco Baiocchi, MD, PhD, Principal Investigator — Department of Gynecologic Oncology - AC Camargo Cancer Center
Locations (5):
- Brazil (5):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital do Cancer de Barretos, Barretos, São Paulo
  - AC Camargo Cancer Center, São Paulo, São Paulo
  - Albert Einstein Hospital, São Paulo, São Paulo
  - Sao Camilo Oncologia, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baiocchi G, Mantoan H, Kumagai LY, Goncalves BT, Badiglian-Filho L, de Oliveira Menezes AN, Faloppa CC, De Brot L, da Costa AABA. The Impact of Sentinel Node-Mapping in Staging High-Risk Endometrial Cancer. Ann Surg Oncol. 2017 Dec;24(13):3981-3987. doi: 10.1245/s10434-017-6132-8. Epub 2017 Oct 20. PMID 29058141
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221
- [Background] Holloway RW, Gupta S, Stavitzski NM, Zhu X, Takimoto EL, Gubbi A, Bigsby GE, Brudie LA, Kendrick JE, Ahmad S. Sentinel lymph node mapping with staging lymphadenectomy for patients with endometrial cancer increases the detection of metastasis. Gynecol Oncol. 2016 May;141(2):206-210. doi: 10.1016/j.ygyno.2016.02.018. Epub 2016 Mar 2. PMID 26905211
- [Background] Soliman PT, Westin SN, Dioun S, Sun CC, Euscher E, Munsell MF, Fleming ND, Levenback C, Frumovitz M, Ramirez PT, Lu KH. A prospective validation study of sentinel lymph node mapping for high-risk endometrial cancer. Gynecol Oncol. 2017 Aug;146(2):234-239. doi: 10.1016/j.ygyno.2017.05.016. Epub 2017 May 18. PMID 28528918
- [Background] Rossi EC, Kowalski LD, Scalici J, Cantrell L, Schuler K, Hanna RK, Method M, Ade M, Ivanova A, Boggess JF. A comparison of sentinel lymph node biopsy to lymphadenectomy for endometrial cancer staging (FIRES trial): a multicentre, prospective, cohort study. Lancet Oncol. 2017 Mar;18(3):384-392. doi: 10.1016/S1470-2045(17)30068-2. Epub 2017 Feb 1. PMID 28159465
- [Background] Bodurtha Smith AJ, Fader AN, Tanner EJ. Sentinel lymph node assessment in endometrial cancer: a systematic review and meta-analysis. Am J Obstet Gynecol. 2017 May;216(5):459-476.e10. doi: 10.1016/j.ajog.2016.11.1033. Epub 2016 Nov 18. PMID 27871836
- [Background] Abu-Rustum NR. Sentinel lymph node mapping for endometrial cancer: a modern approach to surgical staging. J Natl Compr Canc Netw. 2014 Feb;12(2):288-97. doi: 10.6004/jnccn.2014.0026. PMID 24586087
- [Background] Raimond E, Ballester M, Hudry D, Bendifallah S, Darai E, Graesslin O, Coutant C. Impact of sentinel lymph node biopsy on the therapeutic management of early-stage endometrial cancer: Results of a retrospective multicenter study. Gynecol Oncol. 2014 Jun;133(3):506-11. doi: 10.1016/j.ygyno.2014.03.019. Epub 2014 Mar 15. PMID 24642092
- [Derived] Baiocchi G, Andrade CEMC, Ribeiro R, Moretti-Marques R, Tsunoda AT, Alvarenga-Bezerra V, Lopes A, Costa RLR, Kumagai LY, Badiglian-Filho L, Faloppa CC, Mantoan H, De Brot L, Dos Reis R, Goncalves BT. Sentinel lymph node mapping versus sentinel lymph node mapping with systematic lymphadenectomy in endometrial cancer: an open-label, non-inferiority, randomized trial (ALICE trial). Int J Gynecol Cancer. 2022 May 3;32(5):676-679. doi: 10.1136/ijgc-2022-003378. PMID 35236752